CLINICAL TRIAL: NCT01183962
Title: Vitamin D and T-Regulatory Cells in Coronary Artery Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment, funding ended
Sponsor: Creighton University (Other)
Responsible Party: Michael Del Core, MD, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09-15602
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Disease; Cardiovascular Disease
Keywords: CAD; Vitamin D; CVD
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Other): Subject receives daily dose of Vitamin D
  Interventions: Dietary Supplement: Vitamin D
- No medicine (Other): Subject does not receive medication
  Interventions: Other: No medication

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D 3000 IU daily
  Arms: Vitamin D
Other: No medication — No intervention
  Arms: No medicine

SUMMARY:
The purpose of this study is to evaluate the effect of Vitamin D supplementation on cardiovascular disease and certain cells (T-regulatory cells) in the body that play a role in plaque formation in arteries. This study will determine the levels of Vitamin D and T-regulatory cells in subjects with coronary artery disease and if Vitamin D supplementation will affect future events such as heart attach and stroke.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 30 and 80 years
* have a history of medically treated coronary artery disease

Exclusion Criteria:

* history of smoking in the past 2 years
* history of diabetes mellitus

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
increase in T-regulatory Cells | 1 year
  We expect significant improvement in the suppressive capacity, with or without increase in the number, of circulating T-regs after vitamin D supplementation. This increase in T-regs function will correlate with improvement in clinical parameters.

SECONDARY OUTCOMES:
decrease pro-inflammatory cytokines & sTNFR1 and increase serum IL-10 | 1 year
  We also expect that vitamin D supplementation will decrease the levels of pro-inflammatory cytokines and sTNFR1 and increase the level of serum IL-10

CONTACTS AND LOCATIONS:
Overall Officials: Michael DelCore, MD, Principal Investigator — Creighton University
Locations (1):
- The Cardiac Center at Creighton University, Omaha, Nebraska, United States